CLINICAL TRIAL: NCT04267003
Title: Transcranial Direct Current Stimulation (tDCS) Studies of Cognition, Oscillations and GABA Levels in Schizophrenia
Brief Title: Effects of Brain Stimulation on Cognition, Oscillations and GABA Levels in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1515202
Record Dates: First submitted 2020-02-03; First posted 2020-02-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia; EEG; tDCS; dorsolateral prefrontal cortex; cognitive control; transcranial direct current stimulation; GABA; MR spectroscopy
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- DLPFC Stimulation + Task (Experimental): Intervention. 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex during cognitive task completion.
  Interventions: Device: Transcranial Direct Current Stimulation
- DLPFC Stimulation + Rest (Experimental): Intervention. 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex during rest.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Stimulation + Task (Sham Comparator): Placebo Comparator. 0.5-1 minutes of 2 mA direct current stimulation over dorsolateral prefrontal cortex followed by 19-19.5 minutes of sham stimulation, during cognitive task completion.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Stimulation + Rest (Sham Comparator): Placebo Comparator. 0.5-1 minutes of 2 mA direct current stimulation over dorsolateral prefrontal cortex followed by 19-19.5 minutes of sham stimulation, during rest.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, saline-soaked electrodes are temporary affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (~20 minutes) to stimulate the targeted brain area (e.g. the DLPFC). To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation.

SUMMARY:
People with schizophrenia often have problems with attention, learning and memory and other cognitive abilities that interfere with their work and school performance. Unfortunately, even our best treatments often do not significantly reduce these cognitive problems. The current study investigates whether or not delivering a very small electrical current to people's foreheads (called, transcranial direct current stimulation; (tDCS)) might improve functioning in the front part of the brain and reduce these cognitive problems in people with schizophrenia. tDCS is non-invasive and has been shown to improve cognitive functioning in some preliminary studies. The current study will investigate whether giving tDCS during a task is more effective than giving it during rest (Aim 1), whether delivery of tDCS to the front of the head is more effective than delivery to the back of the head (Aim 2), and whether tDCS delivery will alter levels of a major inhibitory neurotransmitter in the brain (GABA; Aim 3) that is important to cognitive functioning and may be disrupted in people with schizophrenia. Although this study is not intended to diagnose, cure or treat schizophrenia or any other disease, if results are positive it will encourage future large-scale studies to determine if tDCS can become an effective treatment for cognitive problems in people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to sufficiently speak and understand English so as to be able to understand and complete cognitive tasks.
* All subjects must have the ability to give valid informed consent.

Inclusion Criteria for Patients with Schizophrenia Only:

* Diagnosis of schizophrenia, schizophreniform or schizoaffective disorder
* No medication changes in the prior month
* No medication changes anticipated in the upcoming month
* Stable outpatient or partial hospital status
* Normal IQ (>70; IQ will be measured by administering the Wechsler Abbreviated Scale of
* Intelligence (WASI) test)
* Must not be currently taking the antipsychotic clozapine

Exclusion Criteria:

* Pacemakers
* Implanted electrical (brain and spinal) stimulators
* Implanted defibrillator
* Metallic implants
* Skin damage or skin conditions such as eczema at the sites where electrodes will be placed
* Hair styles hindering the placement of electrodes
* Cranial pathologies
* Head trauma
* Epilepsy
* Mental retardation
* Any known history of neurological disorders (including epilepsy, amyotrophic lateral sclerosis (ALS), multiple sclerosis (MS), stroke, cerebral palsy, any DSM-5 axis I psychiatric disorder (for healthy control subjects), autism)
* Uncorrected vision problems that would hinder cognitive testing (this also pertains to subjects with color blindness in tasks where discriminating colored objects/items is necessary for successful performance)
* Pregnancy
* Substance dependence in the past six months
* Substance abuse in the past month

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
EEG Correlates of Language and Cognitive Control | Assessment will begin immediately following stimulation and last for about 1.5 hours.
  Electrophysiological data recorded during completion of cognitive control tasks. We will measure oscillatory activity from 3-80 Hz.
Behavioral Response | Assessment will begin immediately following stimulation and last for about 1.5 hours.
  We will assess performance on the Dot Pattern Expectancy (DPX) task (error rates).
Behavioral Response | Assessment will begin immediately following stimulation and last for about 1.5 hours.
  We will assess performance on the Dot Pattern Expectancy (DPX) task (d-prime scores).

CONTACTS AND LOCATIONS:
Locations (1):
- Imaging Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Select data from this study may be submitted to the National Institute of Mental Health Data Archive (NDA). NDA is a data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying mental illness to collect and share de-identified information with each other. The data repository is accessible only to qualified investigators. All subject data will be de-identified (subject names will not be used) and each subject will have a separate identifier called a Global Unique Identifier (GUID) to remove any possibility that "the identities of the subjects cannot be readily ascertained or otherwise associated with the data by the repository staff or secondary data users." (45 CFR, 46.102).

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/effects-of-brain-stimulation-on-cognition-oscillations-and-gaba-levels-in-schizophrenia-205153/